CLINICAL TRIAL: NCT01434199
Title: Does Endoscope Position Detecting Unit Facilitate Caecal Intubation? A Randomized Controlled Trial
Brief Title: Does Endoscope Position Detecting Unit Facilitate a Complete Colonoscopy Examination
Acronym: UPD-3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Sok Fei, Associate consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRE-2011.125-T
Record Dates: First submitted 2011-06-20; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Colorectal Neoplasms
Keywords: magnetic endoscope imaging; colonoscopy; caecal intubation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UPD guided group (Experimental): Both the colonoscopist and assistant will be viewing the imager screen during the whole procedure.
  Interventions: Procedure: UPD guidance
- non-UPD guided group (No Intervention): Conventional colonoscopy would be done without image guidance.

INTERVENTIONS:
Procedure: UPD guidance — A real time, three-dimensional image and position of the colonoscope would be provided to the endoscopist during the procedure.
  Other Names: Magnetic endoscope imaging (MEI)
  Arms: UPD guided group

SUMMARY:
As the incidence of colorectal cancer (CRC) has been rapidly rising in Asian countries, more and more screening colonoscopies are now being performed for prevention or early detection of this fatal disease. Complete colonoscopy as indicated by caecal intubation is essential to make it a reliable screening tool for colorectal cancer or polyps. Cecal intubation rate is highly variable and dependent on individual experience. Colonic looping is the commonest cause of incomplete colonoscopy. Magnetic endoscope imaging (MEI) is a non-radiological imaging technique to provide real time, three-dimensional image and position of the colonoscope during the procedure. It may facilitate straightening of colonic loops and hence cecal intubation.

The investigators aim to evaluate the benefit of MEI in term of cecal intubation rate across endoscopists of all levels of experience by making use of the newly developed Endoscopy Position Detecting Unit (UPD-3)by Olympus Optical Co, Ltd, Japan.

The investigators propose to conduct a prospective randomized controlled trial to compare the caecal intubation rate of colonoscopy being performed with and without UPD-3 guidance. Colonoscopies performed by endoscopists with different level of experience will be randomized to UPD-3 guided group or conventional group (no UPD-3 guidance). Patient controlled sedation (PCS) containing propofol and alfentanil will be given to all patients. The investigators hypothesize that UPD-3 guided colonoscopy is associated with high caecal intubation rate (complete colonoscopy), shorter time to caecum, less patient pain and lower sedative medication requirement. A high caecal intubation rate facilitates a reliable colonoscopy screening. Decreased colonic looping and shorter time to caecum may reduce patient discomfort during the procedure. It may also facilitate learning and acquiring the skill of colonoscopy in trainees.

DETAILED DESCRIPTION:
Hypothesis UPD guided colonoscopy improves cecal intubation rate.

Methods

Trial design This is a prospective randomized controlled trial comparing the cecal intubation rate of colonoscopy being performed with and without UPD guidance by endoscopists of different levels of experience. The trial will be conducted in the Endoscopy Unit of a university affiliated hospital.

Patients who will have elective colonoscopy in the Endoscopy Unit during the study period, and meet the following inclusion criteria are recruited. The colonoscopy will be done by 6 dedicated endoscopists with different levels of experience in performing colonoscopy.

Interventions

UPD-3 and the specific colonoscope with an in-built magnetic imaging facility (Olympus Optical Co, Ltd, Japan) will be used in all examinations. A mobile sensor will be attached to the assistant's hand, so that the hand position in relation to the colonoscope could be shown in the imager screen.

Patient controlled sedation (PCS) will be given to all patients. It is delivered by means of Graseby 3300 PCA pump (Graseby Medical Ltd), using a mixture of propofol (200mg in 20ml) and alfentanil (0.5mg in 1ml) in a 25-ml syringe. The drugs will be delivered in response to pressure on a hand-held button controlled by the patient. Each bolus (0.5ml) delivers 4.8mg propofol and 12microgram alfentanil. No loading dose was used and the lock-out time of the PCA machine was set at zero. All patients will be instructed in the use of the hand-held button before colonoscopy. Nasal oxygen (2l/min) will be given to all patients, and oxygen saturation and blood pressure will be continuously monitored throughout the procedure.

The procedure will be randomized to either with the colonoscopist viewing the imager screen or not.

UPD guided group: Both the colonoscopist and assistant will be viewing the imager screen during the whole procedure. Information about colonoscopy looping will interpreted and documented by the colonoscopist. Anterior-position view is the standard reference. When abdominal compression is required, the assistant nurse should have the hand held probe attached, such that abdominal compression is guided by the image.

Conventional group (non- UPD guided): The imager screen will be turned to the other side such that both the colonoscopist and assistant is blind to UPD images. When the colonoscopist encountered looping as defined by paradoxical movement of the tip or disproportionate advancement in endoscopic view to the shaft insertion, the colonoscopist is requested to estimate the type of loop formed. The images will be captured for later interpretation.

The primary outcome is cecal intubation rate. Cecal intubation is defined as visualization of appendix orifice and ileocaecal valve, procedure started by a trainee and taken over by supervisor before caecal intubation is regarded as incomplete.

Sample size

The cecal intubation rate could be increased by at least 11% for trainee in a randomized trial by Shah [14] and 16% for trainee and experienced endoscopist in another trial [15]. Since the overall cecal intubation rate in our Endoscopy unit without UPD guide is at least 90% already, the investigators expect a modest benefit from UPD guidance. Assume a difference of 5% in caecal intubation rate (from 90% in conventional group to 95% in the UPD guided group) with a power of 80% and a type I error of 5%, 2 sided analysis, 435 patients will be needed in each group. Thus a sample size of 870 patients is required.

Randomization

Informed consent will be obtained before colonoscopy in the Endoscopy Unit, if the patient fulfils the inclusion criteria. Block randomization will be done on a 1:1 basis, to ensure equal number of UPD guided or conventional colonoscopies are done by each endoscopist.

A sealed non-opaque envelope (produced according to the computer generated random sequence) will be opened to determine the appropriate limb of entry before scope insertion.

It is not possible to blind the study.

Statistical analysis

The data will be analyzed according to the intention-to-treat principle. The chi-squared test (or Fisher's exact test when appropriate), Student's t-test, and Mann-Whitney U test will be used to compare categorical, parametric, and non-parametric data, respectively. A P value <0.05 is considered statistically significant.

Planned interim analysis will be conducted after recruiting 50% of patients.

Data collection Data will be collected by the in-charged endoscopist and assistant after each procedure in a standardized data sheet.

Accrual rate It is expected that about 20 cases per week will be recruited for randomization. The study could be finished in around 1 year time.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* American Society of Anaesthesiologist (ASA) grading I-III
* Scheduled for elective colonoscopy

Exclusion Criteria:

* Previous colonic resection
* Refuse to consent to participate
* History of allergy to propofol or alfentanil
* Has a pacemaker in situ
* Pregnant lady

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
caecal intubation rate | 10minutes in average after starting the procedure
  Caeal intubation is the landmark for complete colonoscopy. Caecal intubation would be documented after each procedure. The caecal intubation rate with or without UPD guidance would be compared. The result would provide information whether the UPD device can faciliate complete colonoscopy.

SECONDARY OUTCOMES:
Caecal intubation time | 10 minutes in average after starting the procedure
  Comparison of caecal intubaton time between UPD guided and non-UPD guided group would provide information on whether UPD device faciliate complete colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie SF Hon, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- China (2):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hong Kong
  - Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Shah SG, Brooker JC, Thapar C, Suzuki N, Williams CB, Saunders BP. Effect of magnetic endoscope imaging on patient tolerance and sedation requirements during colonoscopy: a randomized controlled trial. Gastrointest Endosc. 2002 Jun;55(7):832-7. doi: 10.1067/mge.2002.124097. PMID 12024136
- [Background] Shah SG, Brooker JC, Williams CB, Thapar C, Saunders BP. Effect of magnetic endoscope imaging on colonoscopy performance: a randomised controlled trial. Lancet. 2000 Nov 18;356(9243):1718-22. doi: 10.1016/S0140-6736(00)03205-0. PMID 11095259